CLINICAL TRIAL: NCT03357822
Title: A Real-World Study of Sequential Combination Therapy With Pegylated Interferon In Nucleoside-treated Patients With Chronic Hepatitis B
Brief Title: A Real-World Study of Pegylated Interferon In Nucleoside-treated Patients With Chronic Hepatitis B
Acronym: COST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Prof, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COST study
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; Nucleoside analog; Pegylated Interferon; Sequential combination therapy; HBsAg loss
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential combination therapy group (Experimental): Patients are treated with pegylated Interferon (180ug, subcutaneously, once a week) plus entecavir (0.5mg, orally, every day) or tenofovir disoproxil fumarate (300mg, orally, every day) for 48/72/96 weeks
  Interventions: Drug: Pegylated interferon; Drug: Entecavir; Drug: Tenofovir disoproxil fumarate
- Nucleoside therapy group (Active Comparator): Patients are treated with entecavir (0.5mg, orally, every day) or tenofovir disoproxil fumarate (300mg, orally, every day) for 96 weeks
  Interventions: Drug: Entecavir; Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Pegylated interferon — 180ug Pegylated interferon is injected subcutaneously once a week
  Other Names: Pegylated interferon (PegIFN)
  Arms: Sequential combination therapy group
Drug: Entecavir — 0.5mg entecavir is orally taken every day
  Other Names: Entecavir (ETV)
Drug: Tenofovir disoproxil fumarate — 300mg tenofovir is orally taken every day
  Other Names: Tenofovir disoproxil fumarate (TDF)

SUMMARY:
The aim of the prospective real-world study is to evaluate whether sequential combination therapy with pegylated interferon plus entecavir/tenofovir could induce higher rates of HBsAg loss in nucleoside-treated patients with chronic hepatitis B compared to continuous nucleoside treatment.

DETAILED DESCRIPTION:
Patents who were treated with NA at least one year and achieved hepatitis B virus (HBV) DNA suppression and HBsAg level<3000 international unit (IU) /mL are enrolled in this study, they are assigned into two groups, in group I, patients will receive pegylated interferon plus entecavir/tenofovir for 48/72/96 weeks, in group II, patients will receive entecavir/tenofovir for 96 weeks. HBsAg loss rates at the end of treatment and sustained response at the end of follow up will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 18 to 65 years of age;
2. HBsAg positive, entecavir and or adefovir dipivoxil are used at least 1 year including patients with nucleotides or nucleoside resistance history;
3. Before nucleotides or nucleosides treatment, ALT > 2 upper limit of normal value (ULN), HBV DNA >10000 copies/ml, HBsAg positive;
4. Serum HBV DNA ≤ 500 copies/ml;
5. HBsAg<3000 IU/ml;
6. HBsAg positive;
7. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug;
8. Absence of cirrhosis confirmed by ultrasonic test;
9. Agree to participate in the study and sign the patient informed consent.

Exclusion Criteria:

1. HBV DNA > 500 copies/ml;
2. Other antiviral, anti-neoplastic or immunomodulatory treatment (including supra physiologic doses of steroids and radiation) 6 months prior to the first dose of randomized treatment (except for 7 days of acyclovir for herpetic lesions more than 1 month prior to first administration of randomized treatment). Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation are also excluded;
3. Women with ongoing pregnancy or breast-feeding;
4. Co-infection with active hepatitis A, hepatitis C, hepatitis D(Those hospitals which have the ability to do the test will do) and/or human immunodeficiency virus (HIV);
5. ALT >10 ULN;
6. Evidence of decompensated liver disease (Child-Pugh score > 5). Child-Pugh > 5 means, if one of the following 5 conditions are met, the patient has to be excluded:
7. one of the following 5 conditions are met, the patient has to be excluded:
8. Serum albumin < 3.5 g/L;
9. Prothrombin time > 3 seconds prolonged;
10. Serum bilirubin > 34 µ mol/L;
11. History of encephalopathy;
12. History of variceal bleeding;
13. Ascites;
14. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia);
15. Signs or symptoms of hepatocellular carcinoma, patients with a value of alpha-fetoprotein > 100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months. Patients with values < 20 ng/mL but > 100 ng/mL may be enrolled, if hepatic neoplasia has been excluded by liver imaging;
16. Neutrophil count < 1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening;
17. Hemoglobin < 11.5 g/dL for females and <12.5 g/dL for men;
18. Serum creatinine level > 1.5 ULN in screening period.
19. Phosphorus < 0.65 mmol/L;
20. antinuclear antibody (ANA) > 1:100;
21. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease;
22. History of a severe seizure disorder or current anticonvulsant use;
23. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.);
24. History of chronic pulmonary disease associated with functional limitation;
25. Diseases that interferon and nucleotides or nucleosides are not suitable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-01-25 (Estimated); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
HBsAg loss rate | at week 48
  Percentages of patients who achieve HBsAg loss at week 48

SECONDARY OUTCOMES:
HBsAg loss rate | at week 72
  Percentages of patients who achieve HBsAg loss at week 72
HBsAg loss rate | at week 96
  Percentages of patients who achieve HBsAg loss at week 96
HBsAg level | at week 48
  Dynamic change in HBsAg level from baseline to week 48
HBsAg level | at week 72
  Dynamic change in HBsAg level from baseline to week 72
HBsAg level | at week 96
  Dynamic change in HBsAg level from baseline to week 96
sustained HBsAg loss rate | at week 120
  Percentages of patients who achieve HBsAg loss at week 120
decline in HBsAg level | at week 48
  Decline in HBsAg level from baseline to week 48
decline in HBsAg level | at week 72
  Decline in HBsAg level from baseline to week 72
decline in HBsAg level | at week 96
  Decline in HBsAg level from baseline to week 96
HBsAb appearance rate | at week 48
  Percentages of HBsAb appearance at week 48
HBsAb appearance rate | at week 72
  Percentages of HBsAb appearance at week 72
HBsAb appearance rate | at week 96
  Percentages of HBsAb appearance at week 96
HBsAb seroconversion rate | at week 48
  Percentages of HBsAb seroconversion at week 48
HBsAb seroconversion rate | at week 72
  Percentages of HBsAb seroconversion at week 72
HBsAb seroconversion rate | at week 96
  Percentages of HBsAb seroconversion at week 96
HBeAg loss rate | at week 48
  Percentages of HBeAg loss in the HBeAg-positive patients at week 48
HBeAg loss rate | at week 72
  Percentages of HBeAg loss in the HBeAg-positive patients at week 72
HBeAg loss rate | at week 96
  Percentages of HBeAg loss in the HBeAg-positive patients at week 96
HBeAg seroconversion rate | at week 48
  Percentages of HBeAg seroconversion in the HBeAb-negative patients at week 48
HBeAg seroconversion rate | at week 72
  Percentages of HBeAg seroconversion in the HBeAb-negative patients at week 72
HBeAg seroconversion rate | at week 96
  Percentages of HBeAg seroconversion in the HBeAb-negative patients at week 96
Rate of HBV DNA level <1000 copies/mL | at week 96
  Percentages of HBV DNA level <1000 copies/mL at week 96
Rate of alanine aminotransferase (ALT) normalization | at week 96
  Percentages of ALT normalization at week 96
The rate of progression to cirrhosis | at week 120
  The rate of progression to cirrhosis at week 120
The incidence rate of hepatocarcinoma | at week 120
  The incidence rate of hepatocarcinoma at week 120

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, Principal Investigator — Department of Infectious Diseases, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (12):
- China (12):
  - 302 Military Hospital of China, Beijing, Beijing Municipality
  - BeiJing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital Affiliated to AMU, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Zhejiang, Hangzhou
  - Departmen of infectious disease, Xiangya Hospital, Central-south Universit, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Traditional Chinese Medicine,Xiamen Hospital, Shantou, Xiamen
  - The first affiliated hospital of Wenzhou medical universtiy, Wenzhou, Zhejiang